CLINICAL TRIAL: NCT01200459
Title: SMART: A Social and Mobile Weight Control Program for Young Adults
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kevin Patrick, MD, MS, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 090640
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Obesity
Keywords: Obesity; Weight Loss; Healthy Lifestyle; Social; Mobile; Facebook; Text Messages
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Social/Mobile Intervention (Experimental): Theory-based intervention to promote weight loss utilizing web, mobile phone and social media.
  Interventions: Behavioral: Social/mobile weight loss promotion intervention.
- Control (No Intervention): Participants randomized to this group will have access to "usual care" health information via the SMART study website. This arm will be compared to our intervention group.

INTERVENTIONS:
Behavioral: Social/mobile weight loss promotion intervention. — Social/mobile intervention for weight loss promotion, compared to control group.
  Arms: Social/Mobile Intervention

SUMMARY:
The Social/Mobile Approach to Reduce Weight (SMART) study is a 24-month randomized control trial designed to evaluate the hypothesis that weight status at 24 months will be significantly better for the SMART intervention recipients than for those who receive the comparison condition.

DETAILED DESCRIPTION:
The focus of the SMART study is to develop an intervention to promote weight loss in overweight or obese young adults. The investigators will recruit college and university students to evaluate the effects of SMART on weight status and other metabolic, behavioral and psychosocial outcomes up to and including 24 months.

The Primary aim of the study is to evaluate between condition differences in weight status at 24 months.

Secondary aims will assess the impact of the SMART intervention on: Diet, physical activity, sedentary behaviors, quality of life and depression at 6, 12, 18 and 24 months; Anthropometric measures (BP, waist circumference) at 6, 12, 18 and 24 months; Differences in weight status at 6, 18 and 24 months; Level of satisfaction and amount of use of the intervention components.

These aims will be applied to overweight/obese young adults. Among overweight/obese young adults, the investigators will determine whether SMART produces weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 35 years
* Intending to be available for a 24 month intervention
* Full-time student enrollment at one of the designated San Diego college or university campuses: UCSD, SDSU, and CSU San Marcos
* Facebook user or willingness to begin using Facebook
* Owns personal computer
* Owns mobile phone and uses text messaging
* Willing to attend required research measurement visits in San Diego over the 2 year RCT
* Participants must meet overweight and obesity criteria: 25 < BMI <35 kg/m2
* English-speaking
* Able to ambulate unassisted

Exclusion Criteria:

* Those unable to provide informed consent
* Those with a BMI of <25 kg/m2 or >35 kg/m2
* Those who have a household member on the study staff
* Those with any comorbidities of obesity who require immediate sub-specialist referral including pseudo-tumor cerebri, sleep apnea/hypoventilation syndrome, orthopedic problems, and meeting American Diabetes Association criteria for diabetes
* Cardiovascular event within the last 6 months
* Systolic BP at screening of >160 mmHg OR diastolic BP > 100 mmHg
* Current treatment for malignancy other than non-melanoma skin cancer
* Psychiatric or medical condition that prohibit compliance with study protocol, prescribed dietary changes and/or moderate physical activity
* Current treatment for eating disorder
* Taking medications that alter weight
* Regular use of systemic steroids
* Currently pregnant, gave birth within the last 6 months, currently lactating or breastfeeding within the last 3 months or intending to get pregnant over the next two years
* Enrolled in or planning to enroll in another weight loss program
* Past or planned (within the next 24 months) weight loss surgery
* Current participation in a commercial weight loss program
* Investigator discretion
* Non-English speaking
* Not able to ambulate unassisted

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 404 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in weight status | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Godino JG, Merchant G, Norman GJ, Donohue MC, Marshall SJ, Fowler JH, Calfas KJ, Huang JS, Rock CL, Griswold WG, Gupta A, Raab F, Fogg BJ, Robinson TN, Patrick K. Using social and mobile tools for weight loss in overweight and obese young adults (Project SMART): a 2 year, parallel-group, randomised, controlled trial. Lancet Diabetes Endocrinol. 2016 Sep;4(9):747-755. doi: 10.1016/S2213-8587(16)30105-X. Epub 2016 Jul 14. PMID 27426247
- [Derived] Kolodziejczyk JK, Norman GJ, Rock CL, Arredondo EM, Madanat H, Roesch SC, Patrick K. Strategies that predict weight loss among overweight/obese young adults. Am J Health Behav. 2014 Nov;38(6):871-80. doi: 10.5993/AJHB.38.6.9. PMID 25207513
- [Derived] Davila EP, Kolodziejczyk JK, Norman GJ, Calfas K, Huang JS, Rock CL, Griswold W, Fowler JH, Marshall SJ, Gupta A, Patrick K. Relationships between depression, gender, and unhealthy weight loss practices among overweight or obese college students. Eat Behav. 2014 Apr;15(2):271-4. doi: 10.1016/j.eatbeh.2014.03.010. Epub 2014 Mar 27. PMID 24854817
- [Derived] Kolodziejczyk JK, Norman GJ, Roesch SC, Rock CL, Arredondo EM, Madanat H, Patrick K. Exploratory and confirmatory factor analyses and demographic correlate models of the strategies for weight management measure for overweight or obese adults. Am J Health Promot. 2015 Mar-Apr;29(4):e147-57. doi: 10.4278/ajhp.130731-QUAN-391. Epub 2014 Mar 26. PMID 24670075
- [Derived] Patrick K, Marshall SJ, Davila EP, Kolodziejczyk JK, Fowler JH, Calfas KJ, Huang JS, Rock CL, Griswold WG, Gupta A, Merchant G, Norman GJ, Raab F, Donohue MC, Fogg BJ, Robinson TN. Design and implementation of a randomized controlled social and mobile weight loss trial for young adults (project SMART). Contemp Clin Trials. 2014 Jan;37(1):10-8. doi: 10.1016/j.cct.2013.11.001. Epub 2013 Nov 9. PMID 24215774